CLINICAL TRIAL: NCT03992118
Title: Delivering Specialty Care Access Through Use of an Innovative Telehealth-home Based Intervention Feeding Program (Telefeeding) to Address Food Selectivity in Autism Spectrum Disorder
Brief Title: Project LEaH: Learning to Eat at Home
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Holland Bloorview Kids Rehabilitation Hospital (Other)
Responsible Party: Principal Investigator, Sharon Smile, Developmental Paediatrician, Holland Bloorview Kids Rehabilitation Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 18-786
Record Dates: First submitted 2019-06-11; First posted 2019-06-20 (Actual); Last update posted 2020-11-20 (Actual); Status verified 2020-11

CONDITIONS: Autism Spectrum Disorder; Feeding Behavior
MeSH Terms: conditions — Autism Spectrum Disorder; Feeding Behavior

STUDY DESIGN:
Intervention Model Description: Participants will be recruited to participate in a multidisciplinary feeding assessment, after which an intervention plan will be developed to address the participants feeding challenges.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Feeding Challenges (Experimental): Parents will be coached to implement strategies to address factors contributing to feeding challenges based on a multidisciplinary assessment using the medico-oral-behaviour-sensory-environment (MOBSE) approach.
  Interventions: Behavioral: Parent coaching

INTERVENTIONS:
Behavioral: Parent coaching — Parents will be coached to implement behavioural strategies to address factors which are contributing to difficult mealtime behaviours and feeding challenges.

SUMMARY:
The investigators are trying to determine if delivery a feeding intervention program using videoconferencing technology is feasible.

DETAILED DESCRIPTION:
The investigators hope to recruit 10 participants who have a diagnosis of autism spectrum disorder and food selectivity. A Multidisciplinary feeding assessment will be conducted and factors which contribute to the participant's feeding challenges will be identified. Treatment goals will be identified using the Canadian Occupational Performance Measure (COPM). Intervention geared to address the goals identified by parents will be delivered by the clinician(s) via videoconferencing. Participants will participate in up to 12 weekly 1hr visits over the study period.

ELIGIBILITY:
Inclusion Criteria:

* Age: 2-5 years of age
* Diagnosed with Autism Spectrum Disorder
* History of mild to moderate food selectivity
* Access to internet service
* Access to a Windows based laptop with a web camera
* One Parent is available to participate in a 1 hour intervention program within the home environment once per week over a 12 week period.
* English speaking participants
* Parent consents to use of Ontario Telemedicine Network (OTN) technology within in the home.
* Parent is able to use a laptop
* Access to a telephone in order to trouble shoot problems that may arise in setting up OTN technology.

Exclusion Criteria:

* Age: > 6 year of age (rationale being most children will be enrolled in school during the week thus not available for intervention services).

  * History of severe food selectivity
  * No access to internet service and/or laptop
  * History of dysphagia or other swallowing difficulties
  * Oro-motor abnormalities such as cleft lip and palate, macroglossia
  * Presently has a G-tube insitu
  * Participants on medications that may significantly alter appetite such as stimulants and antipsychotic medications.
  * Currently enrolled in a feeding intervention program.

Ages: 2 Years to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 15 (Actual)
Dates: Start 2018-08-07 (Actual); Primary Completion 2020-04-23 (Actual); Study Completion 2020-07-23 (Actual)

PRIMARY OUTCOMES:
Parent Treatment Adherence Scale | 12 weeks
  Parent Treatment Adherence scale will be used to rate parent engagement and understanding of in session materials. The scale will be completed by the therapists at the end of each intervention session to rate parent engagement and understanding of instructions and assignment on a three point likert scale.
Parent Satisfaction Scale | 12 weeks
  A questionnaire was developed for the study to obtain parent feedback at week 12 on the quality of the block of intervention. Questions rated the length of the sessions, number of sessions, the usefulness of teaching tools (for e.g. homework), and participants confidence in handling future feeding challenges. Scores range from 0(strongly disagree) to 4 (strongly agree).
Treatment Fidelity Scale | 12 weeks
  A treatment fidelity checklist was developed for this study. Treatment fidelity will be measured using a questionnaire to rate if the intervention session goals were met during the session. This will be done using a 3 point likert scale. After completion of each session the therapists will rate themselves as: 0= Goal was not achieved; 1- Goal was partially achieved; 2= Goal was fully achieved for each treatment goal for that session.

SECONDARY OUTCOMES:
Change in number of foods eaten from baseline to week 12 (or end of intervention whichever comes first) | 12 weeks
  Number of foods eaten will be captured by a 1 day food diary at baseline and week 12
Change from baseline in performance scores on the COPM scale at 12 weeks | 12 weeks
  Change in participants performance on a single tasks from baseline to 12 weeks (or end of intervention whichever comes first)

CONTACTS AND LOCATIONS:
Overall Officials: Sharon C Smile, MBBS,DM,MSc, Principal Investigator — Holland Bloorview Kids Rehabilitation Hospital
Locations (1):
- Holland Bloorview Kids Rehabilitation Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No